CLINICAL TRIAL: NCT01859663
Title: Baseline Assessment of Dietary Intake and Physical Activity in Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Comparison of Lifestyle Markers Between Women With and Without Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 1303003665
Record Dates: First submitted 2013-05-17; First posted 2013-05-22 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Polycystic Ovary Syndrome; Dietary Habits; Physical Activity
Keywords: Polycystic Ovary Syndrome (PCOS); Diet; Exercise; Questionnaires; Health Beliefs
MeSH Terms: conditions — Polycystic Ovary Syndrome; Feeding Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood and urine samples. Subcutaneous fat biopsy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Women with a past diagnosis of PCOS: We aim to recruit 120 women with a past diagnosis of PCOS. An equal number of lean and overweight/obese women will be recruited within this group based on body mass index (BMI; Lean = 18 - 24 kg/m2 and overweight/obese ≥ 25 kg/m2).
- Women with a history of regular menstrual cycles: We aim to recruit 120 women with a history of regular menstrual cycles. An equal number of lean and overweight/obese women will be recruited within this group based on body mass index (BMI; Lean = 18 - 24 kg/m2 and overweight/obese ≥ 25 kg/m2).
- Women with a history of irregular menstrual cycles: We aim to recruit 120 women with a history of irregular menstrual cycles, and no previous diagnosis of PCOS. An equal number of lean and overweight/obese women will be recruited within this group based on body mass index (BMI; Lean = 18 - 24 kg/m2 and overweight/obese ≥ 25 kg/m2).

SUMMARY:
The purpose of the study is to identify lifestyle factors associated with PCOS and understand how diet and activity levels impact features of PCOS. The secondary aim is to examine psychosocial factors (e.g., health beliefs) of women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is an endocrine disorder that affects 6-12% of reproductive-aged women within the general population. Currently, there is limited knowledge on the current lifestyles of women with PCOS and the psychosocial factors associated with PCOS.

The researchers plan to examine potential lifestyle differences and psychosocial factors between PCOS and healthy women. The Research Team is also interested in the relationships between biological markers and lifestyle endpoints in women with and without PCOS. Previous literature has shown there are biological marker differences between those with and without PCOS. By examining these relationships, researchers may further understand whether PCOS status is associated with lifestyle parameters.

To accomplish these objectives, 360 women (120 women with PCOS, 120 women without PCOS and with normal menstrual cycles, and 120 women without PCOS and with irregular menstrual cycles) will be included in this study. An equal number of lean and overweight/obese women will be recruited within each group based on body mass index (BMI; Lean = 18 - 24 kg/m2 and overweight/obese ≥ 25 kg/m2). Women will be included in the PCOS group if they have a confirmed PCOS diagnosis from their primary care provider. Participants will complete a food frequency questionnaire, a sleep questionnaire, and a physical activity questionnaire. A researcher may also provide participants with a waist-worn accelerometer to monitor physical activity and a wrist-worn accelerometer to monitor sleep for a week. Ultrasound scans of the ovaries will be assessed and the following metabolic parameters will be assessed: (1) 75-gram oral glucose tolerance test; (2) dual X-ray absorptiometry (DXA) scan; (3) vitals and anthropometry assessment to measure waist and hip circumference, height, weight, blood pressure, and heart rate; (4) fasting blood tests to detect androgens (i.e., total testosterone, androstenedione, free androgen index); and (5) an (optional) subcutaneous fat biopsy. Women with and without PCOS will also be asked to complete a questionnaire that will assess the psychosocial factors (e.g., health beliefs). This can be conducted online, in person, or through phone.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 48 years
* BMI ≥ 18 kg/m2
* If ≥ 21 years old, must have completed a pelvic exam in the past 2 years
* In PCOS if: Confirmed PCOS diagnosis from their primary care provider

Exclusion Criteria:

* Use of oral contraceptives, fertility medications, or any drugs known to influence reproductive function
* Pregnant or breastfeeding

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: New York State. Must be between 18-48 years, with a BMI of 18 kg/m2 or higher.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2013-05; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Differences in diet between women with and without PCOS | 1 week
  A food frequency questionnaire will be administered to assess diet composition for the last three months.

SECONDARY OUTCOMES:
Differences in exercise between women with and without PCOS | 1 week
  An accelerometer will be administered to assess physical activity for 1 week.
Differences in psychosocial factors (e.g., health beliefs) of women with and without PCOS | 1-2 weeks
  A questionnaire will be administered to assess psychosocial factors of women with PCOS.
Differences in sleep patterns between women with and without PCOS | 6 consecutive nights
  A wrist-worn accelerometer will be administered to assess sleep patterns for 6 consecutive nights.
LH-FSH ratio | 1 day
  The ratio of circulating LH to FSH concentrations in the serum will be determined for each participant and compared across groups
Hirsutism Score | 1 day
  Degree of hirsutism as judged by the Ferriman-Gallwey scale will be determined and compared across groups
  Degree of hirsutism as judged by the Ferriman-Gallwey scale will be determined and compared across groups
Androgen concentrations | 1 day
  Total testosterone, androstenedione and free androgen index concentrations in serum will be determined and compared across groups.
Menstrual Cycle Length | 1 day
  Average menstrual cycle length as determined by self-reported history will be determined and compared across groups
Body Mass Index | 1 day
  The ratio of weight to height will be determined and compared across groups.
Waist-to-Hip Ratio | 1 day
  The ratio of waist circumference to hip circumference will be determined and compared across groups
Ovarian Volume | 1 day
  The size of each ovary will be determined using ultrasonography for each participant during study participation and compared between groups.
Insulin Sensitivity | 1 day
  Insulin sensitivity will be determined by administration of an oral glucose tolerance test and compared between groups.
Serum progesterone concentration | 1 day
  The serum progesterone concentration will be determined during study participation, assessed in association with luteal dynamics and compared between groups.
Blood pressure | 1 day
  Blood pressure will be determined and compared between groups.
Serum markers of metabolic syndrome | 1 day
  Lipids, glucose and HbA1C concentrations will be determined and compared between groups.
Body fat distribution | 1 day
  Percentage and distribution of fat and lean mass as assessed using DXA technology will be compared between groups.
Subcutaneous fat biopsy (optional) | 1 day
  Subcutaneous fat cells, which represent important sites of reproductive hormone synthesis, will be assessed and compared across groups

CONTACTS AND LOCATIONS:
Overall Officials: Marla E. Lujan, PhD, Principal Investigator — Cornell University
Locations (3):
- United States (3):
  - Human Metabolic Research Unit, Cornell University, Ithaca, New York
  - Strong Fertility Center, Rochester, New York
  - CRC at University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Derived] Lin AW, Dollahite JS, Sobal J, Lujan ME. Health-related knowledge, beliefs and self-efficacy in women with polycystic ovary syndrome. Hum Reprod. 2018 Jan 1;33(1):91-100. doi: 10.1093/humrep/dex351. PMID 29182737